CLINICAL TRIAL: NCT03673462
Title: A Randomized Study to Describe the Safety of an Investigational Quadrivalent Meningococcal Conjugate Vaccine Administered Concomitantly With Routine Pediatric Vaccines in Healthy Infants and Toddlers
Brief Title: Safety of a Quadrivalent Meningococcal Conjugate Vaccine Administered Concomitantly With Routine Pediatric Vaccines in Healthy Infants and Toddlers
Acronym: MET41
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MET41; U1111-1183-6261 (Other: WHO); 2019-004459-35 (EudraCT Number)
Record Dates: First submitted 2018-09-13; First posted 2018-09-17 (Actual); Results first posted 2023-10-05 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Healthy Volunteers (Meningococcal Infection)
MeSH Terms: conditions — Meningococcal Infections | interventions — Meningococcal Vaccines; Tetanus Toxoid; 13-valent pneumococcal vaccine; Rotavirus Vaccines; Hepatitis B Vaccines; Measles-Mumps-Rubella Vaccine; Herpes Zoster Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: A modified double blind design was used. With the exception of the personnel administering the vaccine, everyone involved in study (participants, care provider, investigator, safety outcomes assessor, Sponsor) was blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1: MenACYW Conjugate Vaccine (Experimental): Healthy infants aged greater than equal to (>=) 42 to less than equal to (<=) 89 days (at the time of enrollment) received MenACYW Conjugate Vaccine at the age of Months 2, 4, 6, and 12 along with Pentacel® (DTaP-IPV/Hib vaccine) at 2, 4, and 6 months of age; PREVNAR 13® (pneumococcal 13-valent conjugate vaccine; PCV13) at 2, 4, 6, and 12 months of age; RotaTeq® (rotavirus vaccine) at 2, 4, and 6 months of age; ENGERIX-B® (hepatitis B vaccine) at 2 and 6 months of age; and M-M-R® II (measles, mumps, and rubella vaccine) and VARIVAX® (varicella vaccine) at 12 months of age.
  Interventions: Biological: Meningococcal polysaccharide (serogroups A,C,Y and W) tetanus toxoid Conjugate vaccine (MenACYW Conjugate vaccine); Biological: Diphtheria, Tetanus, Acellular Pertussis, Poliovirus and Haemophilus b Vaccine; Biological: Pneumococcal 13-valent Conjugate Vaccine; Biological: Rotavirus Vaccine; Biological: Hepatitis B Vaccine; Biological: Measles, Mumps, and Rubella Virus Vaccine; Biological: Varicella Virus Vaccine
- Group 2: MENVEO® (Active Comparator): Healthy infants aged >= 42 to <= 89 days (at the time of enrollment) received MENVEO® Conjugate Vaccine at the age of Months 2, 4, 6, and 12 along with Pentacel® (DTaP-IPV/Hib vaccine) at 2, 4, and 6 months of age; PREVNAR 13® (PCV13) at 2, 4, 6, and 12 months of age; RotaTeq® (rotavirus vaccine) at 2, 4, and 6 months of age; ENGERIX-B® (hepatitis B vaccine) at 2 and 6 months of age; and M-M-R® II (measles, mumps, and rubella vaccine) and VARIVAX® (varicella vaccine) at 12 months of age.
  Interventions: Biological: Meningococcal (Groups A, C, Y and W 135) Oligosaccharide Diphtheria CRM197 Conjugate Vaccine (MENVEO®); Biological: Diphtheria, Tetanus, Acellular Pertussis, Poliovirus and Haemophilus b Vaccine; Biological: Pneumococcal 13-valent Conjugate Vaccine; Biological: Rotavirus Vaccine; Biological: Hepatitis B Vaccine; Biological: Measles, Mumps, and Rubella Virus Vaccine; Biological: Varicella Virus Vaccine

INTERVENTIONS:
Biological: Meningococcal polysaccharide (serogroups A,C,Y and W) tetanus toxoid Conjugate vaccine (MenACYW Conjugate vaccine) — Pharmaceutical form: Liquid solution. Route of administration: Intramuscular
  Arms: Group 1: MenACYW Conjugate Vaccine
Biological: Meningococcal (Groups A, C, Y and W 135) Oligosaccharide Diphtheria CRM197 Conjugate Vaccine (MENVEO®) — Pharmaceutical form: Lyophilized powder combined with liquid components Route of administration: Intramuscular
  Arms: Group 2: MENVEO®
Biological: Diphtheria, Tetanus, Acellular Pertussis, Poliovirus and Haemophilus b Vaccine — Pharmaceutical form: Liquid DTaP-IPV to reconstitute lyophilized ActHIB Route of administration: Intramuscular
Biological: Pneumococcal 13-valent Conjugate Vaccine — Pharmaceutical form: Suspension for injection Route of administration: Intramuscular
Biological: Rotavirus Vaccine — Pharmaceutical form: Oral solution Route of administration: Oral
Biological: Hepatitis B Vaccine — Pharmaceutical form: Suspension for injection Route of administration: Intramuscular
Biological: Measles, Mumps, and Rubella Virus Vaccine — Pharmaceutical form: Lyophilized live virus vaccine Route of administration: Subcutaneous
Biological: Varicella Virus Vaccine — Pharmaceutical form: Suspension for injection Route of administration: Subcutaneous

SUMMARY:
The primary objective of this study was to describe the safety profile of Meningococcal Polysaccharide (Serogroups A, C, Y, and W) Tetanus Toxoid (MenACYW) Conjugate Vaccine and Meningococcal (Groups A, C, Y and W 135) Oligosaccharide Diphtheria CRM197 (MENVEO®) Conjugate Vaccine when administered concomitantly with routine pediatric vaccines in healthy infants and toddlers.

DETAILED DESCRIPTION:
Study duration per participant was approximately 16 months, which includes a safety follow-up contact at 6 months after the final vaccination.

ELIGIBILITY:
Inclusion criteria:

* Aged >= 42 to <= 89 days on the day of the first study visit.
* Healthy infants as determined by medical history, physical examination, and judgment of the investigator.
* Informed consent form was signed and dated by the parent(s) or guardian (and by an independent witness if required by local regulations).
* Participant and parent/guardian were able to attend all scheduled visits and complied with all trial procedures.
* Infants who received the first dose of hepatitis B vaccine at least 28 days before the first study visit.

Exclusion criteria:

* Participation at the time of study enrollment or in the 4 weeks preceding the first trial vaccination or planned participation during the present trial period in another clinical trial investigating a vaccine, drug, medical device, or medical procedure.
* Receipt of any vaccine in the 4 weeks preceding the first trial vaccination or planned receipt of any vaccine in the 4 weeks before and / or following any trial vaccination except for influenza vaccination, which might be received at least 2 weeks before or 2 weeks after any study vaccination. This exception includes monovalent pandemic influenza vaccines and multivalent influenza vaccines.
* Previous vaccination against meningococcal disease with either the trial vaccine or another vaccine (i.e., mono- or polyvalent, polysaccharide, or conjugate meningococcal vaccine containing serogroups A, C, Y, or W; or meningococcal B serogroup-containing vaccine).
* Previous vaccination against diphtheria, tetanus, pertussis, poliomyelitis, hepatitis A, measles, mumps, rubella, varicella; and Haemophilus influenzae type b, Streptococcus pneumoniae, and /or rotavirus infection or disease.
* Receipt of more than 1 previous dose of hepatitis B vaccine.
* Receipt of immune globulins, blood or blood-derived products since birth.
* Known or suspected congenital or acquired immunodeficiency; or receipt of immunosuppressive therapy, such as anti-cancer chemotherapy or radiation therapy; or long-term systemic corticosteroid therapy (prednisone or equivalent for more than 2 consecutive weeks) since birth.
* Family history of congenital or hereditary immunodeficiency until the immune competence of the potential vaccine recipient was demonstrated.
* Individuals with blood dyscrasias, leukemia, lymphoma of any type, or other malignant neoplasms affecting the bone marrow or lymphatic systems.
* Individuals with active tuberculosis.
* History of any Neisseria meningitidis infection, confirmed either clinically, serologically, or microbiologically.
* History of diphtheria, tetanus, pertussis, poliomyelitis, hepatitis B, hepatitis A, measles, mumps, rubella, varicella, Haemophilus influenzae type b, Streptococcus pneumoniae, and /or rotavirus infection/disease.
* At high risk for meningococcal infection during the trial (specifically, but not limited to, participants with persistent complement deficiency, with anatomic or functional asplenia, or participants traveling to countries with high endemic or epidemic disease).
* History of intussusception.
* History of any neurologic disorders, including seizures and progressive neurologic disorders.
* History of Guillain-Barré syndrome.
* Known systemic hypersensitivity to any of the vaccine components or to latex, or history of a life-threatening reaction to the vaccine(s) used in the trial or to a vaccine containing any of the same substances, including neomycin, gelatin, and yeast .
* Verbal report of thrombocytopenia contraindicating intramuscular vaccination in the Investigator's opinion.
* Bleeding disorder, or receipt of anticoagulants in the 3 weeks preceding inclusion, contraindicating intramuscular vaccination in the Investigator's opinion.
* Chronic illness (including, but not limited to, cardiac disorders, congenital heart disease, chronic lung disease, renal disorders, auto-immune disorders, diabetes, psychomotor diseases, and known congenital or genetic diseases) that in the opinion of the investigator, is at a stage where it might interfere with trial conduct or completion.
* Any condition which, in the opinion of the Investigator, might interfere with the evaluation of the study objectives.
* Moderate or severe acute illness/infection (according to Investigator judgment) on the day of vaccination or febrile illness (temperature >= 38 degree Celsius [>= 100.4-degree Fahrenheit]). A prospective participant should not be included in the study until the condition has resolved or the febrile event has subsided.
* Identified as a natural or adopted child of the Investigator or employee with direct involvement in the proposed study.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 42 Days to 89 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 2797 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2023-03-16 (Actual); Study Completion 2023-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (69):
- United States (67):
  - Birmingham Pediatric Associates-Site Number:8400049, Birmingham, Alabama
  - Southeastern Pediatric Associates-Site Number:8400034, Dothan, Alabama
  - MedPharmics, LLC - Phoenix-Site Number:8400043, Phoenix, Arizona
  - Northwest Arkansas Pediatric Clinic-Site Number:8400042, Fayetteville, Arkansas
  - HealthStar Research, LLC-Site Number:8400100, Hot Springs, Arkansas
  - The Children's Clinic of Jonesboro, PA-Site Number:8400059, Jonesboro, Arkansas
  - Emmaus Research Center, Inc-Site Number:8400057, Anaheim, California
  - Advanced Clinical Research - Rancho Paseo-Site Number:8400087, Banning, California
  - Premier Health Research Center, LLC-Site Number:8400039, Downey, California
  - Center for Clinical Trials, LLC-Site Number:8400056, Paramount, California
  - Center for Clinical Trials of San Gabriel-Site Number:8400051, West Covina, California
  - Center for Clinical Trials of San Gabriel-Site Number:8400099, West Covina, California
  - Optum Clinical Research-Site Number:8400076, Colorado Springs, Colorado
  - IMMUNOe Research Centers - Thornton-Site Number:8400022, Thornton, Colorado
  - Avail Clinical Research, LLC-Site Number:8400055, DeLand, Florida
  - Advanced Research for Health Improvement-Site Number:8400096, Fort Myers, Florida
  - Sarkis Clinical Trials-Site Number:8400003, Gainesville, Florida
  - De Armas Research Center,-Site Number:8400088, Miami, Florida
  - Healthy Life Research-Site Number:8400075, Miami, Florida
  - Acevedo Clinical Research Associates-Site Number:8400032, Miami, Florida
  - Crystal Biomedical Research-Site Number:8400018, Miami Lakes, Florida
  - Advanced Research for Health Improvement-Site Number:8400005, Naples, Florida
  - Meridian Clinical Research-Site Number:8400114, Macon, Georgia
  - MOC Research-Site Number:8400095, Mishawaka, Indiana
  - Kentucky Pediatics / Adult Research-Site Number:8400044, Bardstown, Kentucky
  - University of Louisville-Site Number:8400082, Louisville, Kentucky
  - Brownsboro Park Pediatrics-Site Number:8400040, Louisville, Kentucky
  - All Children Pediatrics-Site Number:8400069, Louisville, Kentucky
  - MedPharmics-Site Number:8400048, Metairie, Louisiana
  - Pediatric Associates of Fall River-Site Number:8400103, Fall River, Massachusetts
  - MedPharmics Biloxi-Site Number:8400052, Biloxi, Mississippi
  - Craig Spiegel, MD-Site Number:8400067, Bridgeton, Missouri
  - Center for Pharmaceutical Research-Site Number:8400080, Kansas City, Missouri
  - Midwest Childrens Health Research Institute-Site Number:8400060, Lincoln, Nebraska
  - Legacy Pediatrics-Site Number:8400004, Rochester, New York
  - Medication Management-Site Number:8400072, Greensboro, North Carolina
  - Ford, Simpson, Lively & Rice Pediatrics-Site Number:8400021, Winston-Salem, North Carolina
  - Ohio Pediatric Research-Site Number:8400064, Dayton, Ohio
  - PriMed Clinical Research-Site Number:8400033, Dayton, Ohio
  - Senders Pediatrics-Site Number:8400061, South Euclid, Ohio
  - The Children's Center Rehabilitation Hospital-Site Number:8400104, Bethany, Oklahoma
  - Oklahoma State University - Center for Health Sciences-Site Number:8400008, Tulsa, Oklahoma
  - Cyn3rgy Research-Site Number:8400035, Gresham, Oregon
  - Rainbow Pediatrics-Site Number:8400074, Barnwell, South Carolina
  - Coastal Pediatric Research Charleston-Site Number:8400037, Charleston, South Carolina
  - PMG Research of Charleston, LLC-Site Number:8400102, Mt. Pleasant, South Carolina
  - Palmetto Pediatrics, PA-Site Number:8400089, North Charleston, South Carolina
  - PMG Research-Bristol-Site Number:8400009, Bristol, Tennessee
  - Holston Medical Group, Pediatrics at Stone Plaza-Site Number:8400015, Kingsport, Tennessee
  - Pediatric Clinical Trials Tullahoma-Site Number:8400062, Tullahoma, Tennessee
  - ARC Clinical Research at Wilson Parke-Site Number:8400071, Austin, Texas
  - Benchmark Research - Buda-Site Number:8400016, Buda, Texas
  - Crossroads Clinical Research-Site Number:8400058, Corpus Christi, Texas
  - Benchmark Research - San Angelo-Site Number:8400011, San Angelo, Texas
  - Southwest Children's Research Associates, P.A.-Site Number:8400002, San Antonio, Texas
  - Tanner Clinic-Site Number:8400079, Clinton, Utah
  - Wee Care Pediatrics-Site Number:8400065, Kaysville, Utah
  - Murray Pediatrics-Site Number:8400019, Murray, Utah
  - Utah Valley Pediatrics - Timpanogos-Site Number:8400038, Orem, Utah
  - Pediatric Care-Site Number:8400045, Provo, Utah
  - J. Lewis Research-Site Number:8400053, Salt Lake City, Utah
  - Foothill Family Research-South-Site Number:8400036, Salt Lake City, Utah
  - Copperview Medical Center-Site Number:8400068, South Jordan, Utah
  - J Lewis Research Inc-Site Number:8400050, South Jordan, Utah
  - Alliance for Multispecialty Research Syracuse-Site Number:8400066, Syracuse, Utah
  - Pediatric Medical Research of Charlottesville-Site Number:8400077, Charlottesville, Virginia
  - Marshfield Clinic-Site Number:8400054, Marshfield, Wisconsin
- Puerto Rico (2):
  - Investigational Site Number :6300014, San Juan
  - Investigational Site Number :6300108, San Juan

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at 75 sites in Puerto Rico and United States from 17 September 2018 to 16 March 2023.
Pre-assignment Details: A total of 2797 participants were enrolled and randomized in the study.
Period: Overall Study
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: MENVEO®
Started | 2099 | 698
Safety Analysis Set (SafAS) (Safety Analysis Set (SafAS) included all participants who had received at least one dose of the study vaccines and had any safety data available.) | 2080 | 697
Vaccinated at 2 Months | 2080 | 695
Vaccinated at 4 Months | 2005 | 663
Vaccinated at 6 Months | 1951 | 648
Vaccinated at 12 Months | 1838 | 623
Completed | 1799 | 611
Not Completed | 300 | 87
Not completed — Adverse Event | 11 | 1
Not completed — Protocol Violation | 25 | 11
Not completed — Withdrawal by Parent/Guardian | 162 | 56
Not completed — Lost to Follow-up | 102 | 19

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all randomized participants.
Groups:
- Group 1: MenACYW Conjugate Vaccine: Healthy infants aged >= 42 to <= 89 days (at the time of enrollment) received MenACYW Conjugate Vaccine at the age of Months 2, 4, 6, and 12 along with Pentacel® (DTaP-IPV/Hib vaccine) at 2, 4, and 6 months of age; PREVNAR 13® (pneumococcal 13-valent conjugate vaccine; PCV13) at 2, 4, 6, and 12 months of age; RotaTeq® (rotavirus vaccine) at 2, 4, and 6 months of age; ENGERIX-B® (hepatitis B vaccine) at 2 and 6 months of age; and M-M-R® II (measles, mumps, and rubella vaccine) and VARIVAX® (varicella vaccine) at 12 months of age.
- Group 2 MENVEO®: Healthy infants aged >= 42 to <= 89 days (at the time of enrollment) received MENVEO® Conjugate Vaccine at the age of Months 2, 4, 6, and 12 along with Pentacel® (DTaP-IPV/Hib vaccine) at 2, 4, and 6 months of age; PREVNAR 13® (PCV13) at 2, 4, 6, and 12 months of age; RotaTeq® (rotavirus vaccine) at 2, 4, and 6 months of age; ENGERIX-B® (hepatitis B vaccine) at 2 and 6 months of age; and M-M-R® II (measles, mumps, and rubella vaccine) and VARIVAX® (varicella vaccine) at 12 months of age.
- Total: Total of all reporting groups
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2 MENVEO® | Total
Number analyzed (Participants) | 2099 | 698 | 2797
Age, Continuous [Mean (Standard Deviation); unit: days] | 64.7 (6.63) | 64.9 (6.77) | 64.7 (6.67)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 998 | 336 | 1334
  Male | 1101 | 362 | 1463
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 8 | 0 | 8
  Asian | 28 | 12 | 40
  Native Hawaiian or Other Pacific Islander | 10 | 5 | 15
  Black or African American | 210 | 67 | 277
  White | 1719 | 580 | 2299
  More than one race | 102 | 31 | 133
  Unknown or Not Reported | 22 | 3 | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Immediate Unsolicited Systemic Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a clinical investigation participant administered a medicinal product and which did not have any causal relationship with the treatment. An unsolicited AE was an observed AE that did not fulfill the conditions prelisted in the case report book (CRB) in terms of diagnosis and/or onset window post-vaccination. Immediate adverse events are unsolicited systemic adverse events occurring in the 30 minutes after injection. Reported AEs for each arm were presented as pre-specified in protocol.
Time Frame: Within 30 minutes post-any vaccination
Population: Analysis was performed on SafAS that included all participants who had received at least one dose of the study vaccines and had any safety data available.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: MENVEO®
Number analyzed (Participants) | 2080 | 697
Participants | 7 | 2

2. Primary Outcome: Number of Participants With Solicited Injection Site Reactions
Description: A solicited reaction was an "expected" adverse reaction (AR) (sign or symptom) observed and reported under the conditions (nature and onset) pre-listed in the protocol and CRB and considered as related to the product administered. Solicited injection site reactions included Injection site tenderness, Injection site erythema, and Injection site swelling and were planned to be collected and reported for each vaccine separately; and not planned to be collected for Rotavirus vaccine as the vaccine was administered orally, and no injection site reactions were expected to occur. Reported AEs for each arm were presented as pre-specified in protocol.
Time Frame: Within 7 days post any vaccination
Population: Analysis was performed on SafAS. Here, 'Overall number of participants analyzed' = participants with available data for this outcome measure and 'Number analyzed' = participants with available data for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: MENVEO®
Number analyzed (Participants) | 2021 | 676
Participants
  MenACYW or MENVEO: Injection site Tenderness | 1501 | 499
  MenACYW or MENVEO: Injection site Erythema | 826 | 257
  MenACYW or MENVEO: Injection site Swelling: number analyzed (Participants) | 2019 | 676
  MenACYW or MENVEO: Injection site Swelling | 557 | 170
  PENTACEL: Injection site Tenderness: number analyzed (Participants) | 2017 | 676
  PENTACEL: Injection site Tenderness | 1388 | 456
  PENTACEL: Injection site Erythema: number analyzed (Participants) | 2017 | 676
  PENTACEL: Injection site Erythema | 770 | 255
  PENTACEL: Injection site Swelling: number analyzed (Participants) | 2017 | 676
  PENTACEL: Injection site Swelling | 562 | 178
  PREVNAR 13: Injection site Tenderness: number analyzed (Participants) | 2018 | 676
  PREVNAR 13: Injection site Tenderness | 1464 | 496
  PREVNAR 13: Injection site Erythema: number analyzed (Participants) | 2017 | 676
  PREVNAR 13: Injection site Erythema | 889 | 298
  PREVNAR 13: Injection site Swelling: number analyzed (Participants) | 2017 | 676
  PREVNAR 13: Injection site Swelling | 656 | 206
  ENGERIX-B: Injection site Tenderness: number analyzed (Participants) | 2013 | 674
  ENGERIX-B: Injection site Tenderness | 1199 | 395
  ENGERIX-B: Injection site Erythema: number analyzed (Participants) | 2013 | 675
  ENGERIX-B: Injection site Erythema | 539 | 192
  ENGERIX-B: Injection site Swelling: number analyzed (Participants) | 2013 | 675
  ENGERIX-B: Injection site Swelling | 347 | 115
  M-M-R II: Injection site Tenderness: number analyzed (Participants) | 1756 | 588
  M-M-R II: Injection site Tenderness | 786 | 268
  M-M-R II: Injection site Erythema: number analyzed (Participants) | 1755 | 588
  M-M-R II: Injection site Erythema | 409 | 130
  M-M-R II: Injection site Swelling: number analyzed (Participants) | 1754 | 588
  M-M-R II: Injection site Swelling | 221 | 71
  VARIVAX: Injection site Tenderness: number analyzed (Participants) | 1758 | 588
  VARIVAX: Injection site Tenderness | 724 | 252
  VARIVAX: Injection site Erythema: number analyzed (Participants) | 1757 | 588
  VARIVAX: Injection site Erythema | 364 | 129
  VARIVAX: Injection site Swelling: number analyzed (Participants) | 1757 | 588
  VARIVAX: Injection site Swelling | 208 | 70

3. Primary Outcome: Number of Participants With Solicited Systemic Reactions
Description: A solicited reaction was an "expected" AR (sign or symptom) observed and reported under the conditions (nature and onset) pre-listed in the protocol and CRB and considered as related to the product administered. Solicited systemic reactions included fever, vomiting, crying abnormal, drowsiness, appetite loss, and irritability. Reported AEs for each arm were presented as pre-specified in protocol.
Time Frame: Within 7 days post-any vaccination
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: MENVEO®
Number analyzed (Participants) | 2019 | 676
Participants
  Fever: number analyzed (Participants) | 2002 | 671
  Fever | 724 | 219
  Vomiting: number analyzed (Participants) | 2018 | 676
  Vomiting | 542 | 163
  Crying abnormal | 1437 | 478
  Drowsiness: number analyzed (Participants) | 2017 | 676
  Drowsiness | 1430 | 475
  Appetite lost: number analyzed (Participants) | 2018 | 676
  Appetite lost | 1015 | 350
  Irritability: number analyzed (Participants) | 2018 | 676
  Irritability | 1604 | 536

4. Primary Outcome: Number of Participants With Unsolicited Adverse Events
Description: An AE was any untoward medical occurrence in a clinical investigation participant administered a medicinal product, and which does not necessarily have a causal relationship with this treatment. An unsolicited AE was an observed AE that does not fulfill the conditions prelisted in the CRB in terms of diagnosis and/or onset window post-vaccination. Unsolicited AEs includes both serious adverse events (SAEs) and non-serious unsolicited AEs. Reported AEs for each arm were presented as pre-specified in protocol.
Time Frame: Within 30 days post any vaccination
Population: Analysis was performed on SafAS.
Measure: Count of Participants; unit: Participants
Groups:
- Group 1: MenACYW Conjugate Vaccine: Healthy infants aged >= 42 to <= 89 days (at the time of enrollment) received MenACYW Conjugate Vaccine at the age of Months 2, 4, 6, and 12 along with Pentacel® (DTaP-IPV/Hib) at 2, 4, and 6 months of age; PREVNAR 13® (pneumococcal 13-valent conjugate vaccine; PCV13) at 2, 4, 6, and 12 months of age; RotaTeq® (rotavirus vaccine) at 2, 4, and 6 months of age; ENGERIX-B® (hepatitis B vaccine) at 2 and 6 months of age; and M-M-R® II (measles, mumps, and rubella vaccine) and VARIVAX® (varicella vaccine) at 12 months of age.
- Group 2: MENVEO®: Healthy infants aged >= 42 to <= 89 days (at the time of enrollment) received MENVEO® Conjugate Vaccine at the age of Months 2, 4, 6, and 12 along with Pentacel® (DTaP-IPV/Hib) at 2, 4, and 6 months of age; PREVNAR 13® (PCV13) at 2, 4, 6, and 12 months of age; RotaTeq® (rotavirus vaccine) at 2, 4, and 6 months of age; ENGERIX-B® (hepatitis B vaccine) at 2 and 6 months of age; and M-M-R® II (measles, mumps, and rubella vaccine) and VARIVAX® (varicella vaccine) at 12 months of age.
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: MENVEO®
Number analyzed (Participants) | 2080 | 697
Participants | 1352 | 437

5. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs) and Adverse Event of Special Interest (AESIs)
Description: A SAE was any untoward medical occurrence that at any dose resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect, or was an important medical event. An AESI (serious or non-serious) was defined as one of scientific and medical concern specific to the Sponsor's product or program, for which ongoing monitoring and rapid communication by the Investigator to the Sponsor was appropriate. Reported AEs for each arm were presented as pre-specified in protocol.
Time Frame: From day of first vaccination (i.e., at the age of 2 months) up to 6 months after last vaccination (i.e., up to the age of 18 months)
Population: Analysis was performed on SafAS.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: MENVEO®
Number analyzed (Participants) | 2080 | 697
Participants
  SAE | 108 | 21
  AESI | 19 | 1

6. Primary Outcome: Number of Participants With Medically Attended Adverse Event (MAAEs)
Description: A MAAE was defined as a new onset of a condition that prompts the participant or participant's parent/guardian to seek unplanned medical advice at a health care provider's office or Emergency Department. Reported AEs for each arm were presented as pre-specified in protocol.
Time Frame: as for outcome 5
Population: Analysis was performed on SafAS.
Measure: Count of Participants; unit: Participants
Groups:
- MENVEO®: Healthy infants aged >= 42 to <= 89 days (at the time of enrollment) received MENVEO® Conjugate Vaccine at the age of Months 2, 4, 6, and 12 along with Pentacel® (DTaP-IPV/Hib) at 2, 4, and 6 months of age; PREVNAR 13® (PCV13) at 2, 4, 6, and 12 months of age; RotaTeq® (rotavirus vaccine) at 2, 4, and 6 months of age; ENGERIX-B® (hepatitis B vaccine) at 2 and 6 months of age; and M-M-R® II (measles, mumps, and rubella vaccine) and VARIVAX® (varicella vaccine) at 12 months of age.
Arm/Group | Group 1: MenACYW Conjugate Vaccine | MENVEO®
Number analyzed (Participants) | 2080 | 697
Participants | 1581 | 526

ADVERSE EVENTS:
Time Frame: Unsolicited AE: within 30 days post-any vaccination. Solicited Reactions (SR): within 7 days post-any vaccination. SAE: from day of first vaccination (i.e., at the age of 2 months) up to 6 months post last vaccination (i.e., up to the age of 18 months)
Description: Solicited reaction was an "expected" AR (sign or symptom) observed & reported under conditions (nature & onset) pre-listed in the protocol and CRB. Unsolicited AE: observed AE that does not fulfill the conditions prelisted in the CRB. SafAS. Reported AEs for each arm were presented as pre-specified in protocol. In AE section, solicited reactions fever, crying abnormal, drowsiness, and appetite lost are reported under Pyrexia, crying, somnolence, and decreased appetite, respectively.
Groups:
- Group 2: MENVEO®: Healthy infants aged >= 42 to <= 89 days (at the time of enrollment) received MENVEO® Conjugate Vaccine at the age of Months 2, 4, 6, and 12 along with Pentacel® (DTaP-IPV//Hib) at 2, 4, and 6 months of age; PREVNAR 13® (PCV13) at 2, 4, 6, and 12 months of age; RotaTeq® (rotavirus vaccine) at 2, 4, and 6 months of age; ENGERIX-B® (hepatitis B vaccine) at 2 and 6 months of age; and M-M-R® II (measles, mumps, and rubella vaccine) and VARIVAX® (varicella vaccine) at 12 months of age.
Arm/Group | Group 1: MenACYW Conjugate Vaccine | Group 2: MENVEO®
All-Cause Mortality (participants affected / at risk) | 3/2080 | 0/697
Serious Adverse Events (participants affected / at risk) | 108/2080 | 21/697
Other Adverse Events (participants affected / at risk) | 1889/2080 | 642/697
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: MenACYW Conjugate Vaccine (N=2080) | Group 2: MENVEO® (N=697)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Alagille Syndrome (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Congenital Absence Of Bile Ducts (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Craniosynostosis (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Laryngomalacia (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Bowel Movement Irregularity (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastroenteritis Eosinophilic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 3 (3) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Incarcerated Inguinal Hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intussusception (Gastrointestinal disorders) | 1 (1) | 0 (0)
Necrotising Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Sandifer's Syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Developmental Delay (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 2 (4) | 0 (0)
Sudden Infant Death Syndrome (General disorders) | 1 (1) | 0 (0)
Anaphylactic Reaction (Immune system disorders) | 1 (1) | 0 (0)
Acinetobacter Infection (Infections and infestations) | 1 (1) | 0 (0)
Adenoviral Upper Respiratory Infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 9 (9) | 1 (1)
Covid-19 (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis Orbital (Infections and infestations) | 1 (1) | 0 (0)
Croup Infectious (Infections and infestations) | 0 (0) | 2 (2)
Epstein-Barr Virus Infection (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis Viral (Infections and infestations) | 4 (4) | 0 (0)
Hand-Foot-And-Mouth Disease (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Mastoiditis (Infections and infestations) | 1 (1) | 0 (0)
Metapneumovirus Bronchiolitis (Infections and infestations) | 1 (1) | 0 (0)
Parainfluenzae Virus Infection (Infections and infestations) | 0 (0) | 1 (1)
Perineal Abscess (Infections and infestations) | 0 (0) | 1 (1)
Pharyngeal Abscess (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 1 (2)
Respiratory Syncytial Virus Bronchiolitis (Infections and infestations) | 7 (7) | 1 (1)
Respiratory Syncytial Virus Infection (Infections and infestations) | 11 (11) | 1 (1)
Rhinovirus Infection (Infections and infestations) | 2 (2) | 2 (2)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Septic Shock (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal Scalded Skin Syndrome (Infections and infestations) | 1 (1) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 3 (3) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 0 (0)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0)
Wound Infection (Infections and infestations) | 1 (1) | 0 (0)
Accidental Exposure To Product (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Extradural Haematoma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Head Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Multiple Fractures (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skull Fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Subdural Haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Thermal Burn (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Hepatic Enzyme Increased (Investigations) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 5 (5) | 3 (3)
Failure To Thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Metabolic Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Adrenocortical Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Epilepsy (Nervous system disorders) | 2 (2) | 0 (0)
Febrile Convulsion (Nervous system disorders) | 15 (16) | 1 (1)
Fontanelle Bulging (Nervous system disorders) | 1 (1) | 0 (0)
Haemorrhage Intracranial (Nervous system disorders) | 1 (1) | 0 (0)
Hypotonia (Nervous system disorders) | 1 (1) | 0 (0)
Loss Of Consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 3 (3) | 1 (1)
Seizure Like Phenomena (Nervous system disorders) | 1 (1) | 0 (0)
Unresponsive To Stimuli (Nervous system disorders) | 1 (1) | 0 (0)
Mental Status Changes (Psychiatric disorders) | 2 (2) | 0 (0)
Stereotypy (Psychiatric disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchial Hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: MenACYW Conjugate Vaccine (N=2080) | Group 2: MENVEO® (N=697)
Diarrhoea (Gastrointestinal disorders) | 85 (92) | 37 (39)
Teething (Gastrointestinal disorders) | 161 (200) | 60 (68)
Vomiting (Gastrointestinal disorders) | 579 (807) | 172 (253)
Crying (General disorders) | 1439 (3327) | 479 (1125)
Injection Site Bruising (General disorders) | 353 (742) | 107 (223)
Injection Site Erythema (General disorders) | 1129 (6150) | 380 (2025)
Injection Site Pain (General disorders) | 1619 (13051) | 538 (4340)
Injection Site Swelling (General disorders) | 871 (3790) | 282 (1196)
Pyrexia (General disorders) | 810 (1280) | 248 (360)
Otitis Media (Infections and infestations) | 148 (176) | 47 (56)
Otitis Media Acute (Infections and infestations) | 106 (132) | 30 (34)
Upper Respiratory Tract Infection (Infections and infestations) | 297 (340) | 89 (99)
Decreased Appetite (Metabolism and nutrition disorders) | 1017 (1857) | 351 (611)
Somnolence (Nervous system disorders) | 1430 (3462) | 475 (1127)
Irritability (Psychiatric disorders) | 1604 (4314) | 538 (1476)
Cough (Respiratory, thoracic and mediastinal disorders) | 105 (113) | 30 (31)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable participant matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.

DOCUMENTS (2):
  • Study Protocol (2019-05-29): https://cdn.clinicaltrials.gov/large-docs/62/NCT03673462/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-15): https://cdn.clinicaltrials.gov/large-docs/62/NCT03673462/SAP_001.pdf